CLINICAL TRIAL: NCT05148949
Title: Safety and Immunogenicity of Three Doses of an Inactivated SARS-CoV-2 Vaccine in Chinese Pulmonary Tuberculosis Patients Aged 18-75 Years: a Randomized, Double-blind, Parallel-controlled Clinical Trial
Brief Title: Study on Three Doses of an Inactivated COVID-19 Vaccine in Chinese Pulmonary Tuberculosis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT134
Record Dates: First submitted 2021-12-03; First posted 2021-12-08 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2021-12

CONDITIONS: COVID-19; Pulmonary Tuberculosis
MeSH Terms: conditions — COVID-19; Tuberculosis, Pulmonary

STUDY DESIGN:
Intervention Model Description: Pulmonary tuberculosis patients will be randomized at a 1:1 ratio to receive two doses of standard dosage CoronaVac plus one dose of double dosage CoronaVac or two doses of standard dosage CoronaVac plus one dose of standard dosage CoronaVac at a schedule of 0, 28, 56 days, respectively. Healthy subjects served as an external control group will be vaccinated with two doses of standard dosage CoronaVac at a schedule of 0, 28 days.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and investigators will be kept blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Investigational vaccine group 1 (Experimental): 100 tuberculosis patients will receive two doses of standard dosage CoronaVac plus one dose of double dosage CoronaVac at a schedule of 0, 28, 56 days.
  Interventions: Biological: Standard dosage inactivated vaccine; Biological: Double dosage inactivated vaccine
- Investigational vaccine group 2 (Experimental): 100 tuberculosis patients will receive two doses of standard dosage CoronaVac plus one dose of standard dosage CoronaVac at a schedule of 0, 28, 56 days.
  Interventions: Biological: Standard dosage inactivated vaccine; Biological: Double dosage inactivated vaccine
- Standard regimen group (Active Comparator): 40 healthy subjects will receive two doses of standard dosage CoronaVac at a schedule of 0, 28 days.
  Interventions: Biological: Standard dosage inactivated vaccine

INTERVENTIONS:
Biological: Standard dosage inactivated vaccine — This vaccine contains 600 SU of SARS-CoV-2 antigen, which is produced by Sinovac Research & Development Co., Ltd. 0.5 ml / bottle.
  Other Names: Standard dosage CoronaVac
Biological: Double dosage inactivated vaccine — This vaccine contains 1200 SU of SARS-CoV-2 antigen, which is produced by Sinovac Research & Development Co., Ltd. 0.5 ml / bottle.
  Other Names: Double dosage CoronaVac
  Arms: Investigational vaccine group 1; Investigational vaccine group 2

SUMMARY:
This is a randomized, double-blind, parallel-controlled study, for evaluation of safety and immunogenicity of three doses of an inactivated COVID-19 vaccine (CoronaVac) in pulmonary tuberculosis patients aged 18-75 years. 200 tuberculosis patients and 40 healthy adults aged 18-75 years will be recruited in this study. Of them, 200 pulmonary tuberculosis patients will be randomized at a 1:1 ratio to receive two doses of standard dosage CoronaVac plus one dose of double dosage CoronaVac or two doses of standard dosage CoronaVac plus one dose of standard dosage CoronaVac at a schedule of 0, 28, 56 days, respectively. Other 40 healthy subjects served as an external control group will be vaccinated with two doses of standard dosage CoronaVac at a schedule of 0, 28 days. The occurrence of adverse events within 28 days after each dose vaccination and serious adverse events within 3 months after full vaccination will be observed. In addition, blood samples will be collected on day 0 before the first dose and 28 days and 3 months after the last dose vaccination in all participants and 28 days after second dose in pulmonary tuberculosis patients. Each subject will remain in this study for 5 months (healthy group) or 6 months (tuberculosis group).

ELIGIBILITY:
Inclusion criteria for pulmonary tuberculosis patients:

1. Pulmonary tuberculosis patients aged 18-75 years who have not received COVID-19 vaccine.
2. The condition is determined to be stable by the clinician.
3. The subjects can provide with informed consent and sign informed consent form (ICF).
4. The subjects are able to and willing to comply with the requirements of the clinical trial program and could complete the follow-up of the study.
5. Axillary temperature ≤ 37.0℃.

Inclusion criteria for healthy participants:

1.Healthy subjects aged 18-75 years who have not received COVID-19 vaccine. 2.The subjects can provide with informed consent and sign informed consent form (ICF).

3.The subjects are able to and willing to comply with the requirements of the clinical trial program and could complete the follow-up of the study.

4.Axillary temperature ≤ 37.0℃. Exclusion criteria for the first vaccination

1. Medical history or family history of convulsion, epilepsy, encephalopathy and psychosis.
2. HIV positive.
3. Cancer patients under treatment.
4. Allergic to any component of the research vaccines, or a history of hypersensitivity or serious reactions to vaccination.
5. Women with positive urine pregnancy test, pregnant or breast-feeding, or have a pregnancy plan in this study.
6. Severe chronic diseases or condition in progress cannot be controlled.( Grade 3 or higher as defined in the guidelines for the classification of adverse events in clinical trials for prophylactic vaccines).
7. Transaminase ≥ 3 times ULN or total bilirubin ≥2 times ULN, or other serious adverse reactions as determined by the clinician for antituberculosis treatment.
8. Congenital or acquired angioedema / neuroedema.
9. Asplenia or functional asplenia.
10. Thrombocytopenia or other clotting disorder (this may contraindicate intramuscular injection).
11. Immunosuppressant therapy, antiallergic therapy, cytotoxic therapy, high dose inhaled corticosteroid over the past 6 months (excluding corticosteroid spray for allergic rhinitis, surface corticosteroid for acute non-complicated dermatitis, and corticosteroid with dose less than 20mg/ day)
12. Received blood products within 4 months before vaccination.
13. Received other investigational drugs within 1 month prior to receiving the investigational vaccines.
14. Received other live attenuated vaccines within 1 month prior to receiving the investigational vaccines.
15. Received subunit or inactivated vaccine within 14 days prior to receiving investigational vaccine.
16. Any medical, psychological, social or other conditions that, in the investigator's judgment, are inconsistent with the study protocol or affect the subjects' informed consent Exclusion criteria for subsequent vaccination

1.Those who have had a severe allergic reaction after a previous dose of vaccine.

2.Serious adverse events causally related to the previous vaccination. 3.The newly discovered or newly emerging cases who don't meet the inclusion criteria or meet the exclusion criteria for the first dose, the investigator will decide whether they will continue to participate in the study.

4.Other reasons the investigator consider for exclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-03-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse reaction within 28 days after each dose | within 28 days after each dose
  Incidence of adverse reaction within 28 days after each dose.
GMT of neutralizing antibodies against live SARS-CoV-2 virus on day 28 after the second dose. | On day 28 after the second dose
  GMT of neutralizing antibodies against live SARS-CoV-2 virus on day 28 after the second dose.

SECONDARY OUTCOMES:
Incidence of solicited adverse events within 7 days after each dose. | within 7 days after each dose
  Incidence of solicited adverse events within 7 days after each dose.
Incidence of adverse events within 28 days after each dose. | within 28 days after each dose
  Incidence of adverse events within 28 days after each dose.
Incidence of unsolicited adverse events within 28 days after each dose. | within 28 days after each dose
  Incidence of unsolicited adverse events within 28 days after each dose.
Incidence of serious adverse events (SAE) till the 3 months after the last vaccination. | within 3 months after the last vaccination
  Incidence of serious adverse events (SAE) till the 3 months after the last vaccination.
GMT of anti-S protein of SARS-CoV-2 binding antibodies on day 28 and month 3 after the last dose in all groups and day 28 after second dose in pulmonary tuberculosis patients. | on day 28 and month 3 after the last dose in all groups and day 28 after second dose in pulmonary tuberculosis patients
  GMT of anti-S protein of SARS-CoV-2 binding antibodies measured by ELISA on day 28 and month 3 after the last dose in all groups and day 28 after second dose in tuberculosis patients.
Fold increase of anti-S protein of SARS-CoV-2 binding antibodies on day 28 and month 3 after the last dose in all groups and day 28 after second dose in pulmonary tuberculosis patients. | on day 28 and month 3 after the last dose in all groups and day 28 after second dose in pulmonary tuberculosis patients
  Fold increase of anti-S protein of SARS-CoV-2 binding antibodies on day 28 and month 3 after the last dose in all groups and day 28 after second dose in pulmonary tuberculosis patients.
GMT of neutralizing antibodies against live SARS-CoV-2 virus on day 28 and month 3 after the last dose in pulmonary tuberculosis patients. | on day 28 and month 3 after the last dose in pulmonary tuberculosis patients
  GMT of neutralizing antibodies against live SARS-CoV-2 virus on day 28 and month 3 after the last dose in pulmonary tuberculosis patients.
8. Fold increase of neutralizing antibodies against live SARS-CoV-2 virus on day 28 and month 3 after the last dose in all groups and day 28 after second dose in pulmonary tuberculosis patients. | on day 28 and month 3 after the last dose in all groups and day 28 after second dose in pulmonary tuberculosis patients
  Fold increase of neutralizing antibodies against live SARS-CoV-2 virus on day 28 and month 3 after the last dose in all groups and day 28 after second dose in pulmonary tuberculosis patients.

OTHER OUTCOMES:
GMT of neutralizing antibodies against SARS-CoV-2 variants on day 28 and month 3 after the last dose in all groups and day 28 after second dose in pulmonary tuberculosis patients. | on day 28 and month 3 after the last dose in all groups and day 28 after second dose in pulmonary tuberculosis patients
  GMT of neutralizing antibodies against SARS-CoV-2 variants on day 28 and month 3 after the last dose in all groups and day 28 after second dose in pulmonary tuberculosis patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Xin Li, PhD, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention; Li-mei Zhu, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (6):
- China (6):
  - Huai'an No.4 People's Hospital, Huai'an, Jiangsu
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - Wuxi No.5 People's Hospital, Wuxi, Jiangsu
  - Xuzhou Infectious Disease Hospital, Xuzhou, Jiangsu
  - Binhai County Hospital of Chinese medicine, Yancheng, Jiangsu
  - Danyang Center for Disease Control and Prevention, Zhenjiang, Jiangsu

REFERENCES:
- [Derived] Jin P, Liu Q, Chen W, Guo X, Jiang H, Zhang R, Ding M, Zhang K, Cao Z, He J, Jia S, Wei M, Hu Y, Cui L, Wang J, Li Z, Zhang X, Xia X, Wu Y, Zhou L, Zhu Y, Gao C, Zhang T, Zhu F, Zeng G, Zhu L, Li J. Immunogenicity and safety of two-dose or three-dose regimens of inactivated COVID-19 vaccines in patients with pulmonary tuberculosis: a randomised clinical trial. Expert Rev Vaccines. 2024 Jan-Dec;23(1):1041-1051. doi: 10.1080/14760584.2024.2425283. Epub 2024 Nov 11. PMID 39523878